CLINICAL TRIAL: NCT01049906
Title: A Study to Determine the Quality of Sensory and Motor Blockade of Popliteal Sciatic Nerve Block Catheters Placed Under Ultrasound Guidance With and Without Nerve Stimulation
Brief Title: Popliteal Sciatic Nerve Block Catheter Placement for Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Christopher Robards, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07-008192
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Foot Surgery; Ankle Surgery
Keywords: foot surgery; ankle surgery; Patients scheduled for foot and ankle surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve stimulation and Ultrasound (Active Comparator)
  Interventions: Procedure: Placement of nerve block catheter
- Ultrasound without nerve stimulation (Active Comparator)
  Interventions: Procedure: Placement of nerve block catheter

INTERVENTIONS:
Procedure: Placement of nerve block catheter — Placement of nerve block catheter with nerve stimulator and ultrasound
  Arms: Nerve stimulation and Ultrasound
Procedure: Placement of nerve block catheter — Placement of nerve block catheter with ultrasound only
  Arms: Ultrasound without nerve stimulation

SUMMARY:
Hypothesis: When performed under ultrasound guidance, there is improvement in the sensory and motor blockade obtained with stimulating popliteal catheters versus those placed without nerve stimulation.

ELIGIBILITY:
Inclusion criteria:

* patients scheduled to undergo foot or ankle surgery at Mayo Clinic Jacksonville

Exclusion criteria:

* emergency surgery
* peripheral neuropathy in the distribution of the sciatic nerve on the operative side
* history of recent alcohol or drug abuse
* allergy to local anesthetics
* pregnancy
* coagulopathy
* subjects declined to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complete motor and sensory anesthesia in the sciatic nerve distribution. | Upon block placement

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Robards, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States